CLINICAL TRIAL: NCT04937634
Title: Pharmacokinetic Study of Melphalan in Pediatric Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Food and Drug Safety Evaluation (Republic of Korea) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-MIDD-Mel
Record Dates: First submitted 2021-03-28; First posted 2021-06-24 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Melphalan; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Melphalan (Experimental)
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — The subject receives conditioning regimen including melphalan as a part of hematopoietic stem cell transplantation. Dosage of melphalan is 50mg/m^2/day. Infuse Melphalan over 30 minutes.
  Other Names: Conditioning regimen including melphalan for hematopoietic stem cell transplantation

SUMMARY:
This is an investigator-initiated clinical trial to analysis melphalan pharmacokinetics in pediatric hematopoietic stem cell transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient who will receive a conditioning regimen including melphalan as a part of hematopoietic stem cell transplantation (HSCT).
* Age is below 19 at the time of diagnosis of a disease which is HSCT indication
* Written Study Informed consent and/or assent from the patient, parent, or guardian

Exclusion Criteria:

* Female patients who are pregnant or breast feeding
* Study treatment would deteriorate patient's disease.
* The patient may have problems with study participation due to a psychotic disorder.
* Any condition that would, in the Investigator's judgement, interfere with participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Melphalan concentration | pre dose, within 5 minutes from end of melphalan infusion(EOI), 40 minutes from EOI, 70 minutes from EOI, 170 minutes from EOI
  Analysis: Maximum Concentration observed (Cmax)
Melphalan concentration | pre dose, within 5 minutes from end of melphalan infusion(EOI), 40 minutes from EOI, 70 minutes from EOI, 170 minutes from EOI
  Analysis: Time of Maximum concentration observed (Tmax)
Melphalan concentration | pre dose, within 5 minutes from end of melphalan infusion(EOI), 40 minutes from EOI, 70 minutes from EOI, 170 minutes from EOI
  Analysis: Area Under the Curve
Melphalan concentration | pre dose, within 5 minutes from end of melphalan infusion(EOI), 40 minutes from EOI, 70 minutes from EOI, 170 minutes from EOI
  Analysis: Half lite (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea